CLINICAL TRIAL: NCT01637467
Title: The Effects of Electrical Muscle Stimulation (EMS) on Muscle Atrophy and Functional Outcomes in Critically Ill Patients; a Pilot Randomized Controlled Trial
Brief Title: Effect of Electrical Muscle Stimulation in Critically Ill Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Lung Association (Unknown)
Responsible Party: Principal Investigator, Sunita Mathur, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0639A
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2015-05

CONDITIONS: Critical Illness
Keywords: critical illness; myopathy; electrical muscle stimulation
MeSH Terms: conditions — Critical Illness; Muscular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMS intervention (Experimental): The experimental group will received EMS at a therapeutic level.
  Interventions: Other: Electrical muscle stimulation (EMS)
- Sham (Sham Comparator): The sham group will receive EMS at a sub-therapeutic level.
  Interventions: Other: Sham EMS

INTERVENTIONS:
Other: Electrical muscle stimulation (EMS) — EMS delivered to the quadriceps and gluteal muscles, twice daily, 30 minutes per session for up to 4 weeks.
  Arms: EMS intervention
Other: Sham EMS — Sham EMS delivered to the quadriceps and gluteal muscles, twice daily, 30 minutes per session for up to 4 weeks.
  Arms: Sham

SUMMARY:
Electrical muscle stimulation (EMS) is the therapy used to passively activate muscles using electrodes on the surface of the skin. EMS may be helpful in preserving muscle function in people who are on bedrest due to critical illness in the intensive care unit. The purpose of this study is to determine the safety and feasibility of implementing EMS in critically ill patients who are on mechanical ventilation for greater than 7 days, and examine the effects of 4 weeks of EMS on leg muscle size, muscle strength and functional outcomes in these patients. The investigators hypothesize that EMS will be safe and feasible and that critically ill patients receiving EMS will show a smaller loss of muscle size and strength than those in the control group, who do not receive EMS.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the medical-surgical ICU or cardiovascular ICU
* walking independently prior to admission
* mechanically ventilated for more than 7 days (i.e. prolonged ventilation)
* receiving enteral or parenteral nutrition.

Exclusion Criteria:

* history of neurological or psychiatric disease
* primary muscle disease (e.g. muscular dystrophy, polymyositis)
* catastrophic neurological event
* receiving palliative care
* contraindications to EMS (e.g. cardiac pacemaker/defibrillator, pregnancy, infected or cancerous lesions in proximity of electrode sites)
* inadequate access to electrode sites due to medical devices
* lower extremity edema affecting the thighs or buttocks
* BMI > 35 kg/m2
* allergies to adhesives or latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
feasibility of EMS treatment | 4 weeks
  the number of EMS treatments that are successfully applied will be expressed as a frequency of the total number of treatments attempted

SECONDARY OUTCOMES:
muscle strength | baseline, 2 weeks and 4 weeks
  muscle strength using manual muscle testing
muscle thickness | baseline, 2 weeks, 4 weeks
  thickness of the quadriceps muscle will be assessed using muscle ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lo, BSc(PT), Principal Investigator — University Health Network, Toronto; Sunita Mathur, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada